CLINICAL TRIAL: NCT07274644
Title: Effects of iGlarLixi Versus iGlar on Liver Fat Content in Patients With Type 2 Diabetes Mellitus With Metabolic Dysfunction-associated Steatotic Liver Disease: A Randomized Controlled Trial
Brief Title: Effects of iGlarLixi Versus iGlar on Liver Fat Content in Patients With Type 2 Diabetes Mellitus Combined With Metabolic Dysfunction-associated Steatotic Liver Disease
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Yan Bi, Chief Physician, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-325-03
Record Dates: First submitted 2025-11-24; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-03

CONDITIONS: Metabolic Dysfunction-Associated Steatotic Liver Disease; Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iGlarLixi group (Experimental): Participants receive iGlarLixi once daily before breakfast for 12 weeks.
  Interventions: Drug: iGlarLixi
- iGlar group (Other): Participants receive iGlar once daily at a fixed time for 12 weeks.
  Interventions: Drug: IGlar U100

INTERVENTIONS:
Drug: iGlarLixi — The iGlarLixi is administered as a subcutaneous injection once daily within 1 hour before breakfast. The starting dose ranges from 0.1 to 0.2 U/kg, with a maximum daily dose of 20 U (equivalent to 20 U iGlar or 20 μg Lixi). Dose titration is guided by fasting self-monitored plasma glucose (SMPG) levels, with the goal of achieving a target range of 4.4-5.6 mmol/L while avoiding hypoglycemia. All participants continue to receive background metformin therapy throughout the treatment period.
  Arms: iGlarLixi group
Drug: IGlar U100 — The iGlar is administered via subcutaneous injection once daily at a fixed time. The recommended starting dose ranges from 0.1 to 0.2 U/kg. The dose is subsequently titrated to achieve a fasting self-monitored plasma glucose (SMPG) target of 4.4-5.6 mmol/L, with careful attention to avoiding hypoglycemia. Throughout the study, all participants maintain their background metformin therapy
  Arms: iGlar group

SUMMARY:
This is a single-center, randomized, open-label, controlled clinical trial to compare the effects of a fixed-ratio combination of insulin glargine 100 U/mL plus lixisenatide (iGlarLixi) versus insulin glargine 100 U/mL (iGlar) on liver fat content in patients with Type 2 Diabetes (T2DM) and Metabolic Dysfunction-Associated Steatotic Liver Disease (MASLD). The study includes a 12-week treatment period.

DETAILED DESCRIPTION:
This study is designed as a single-center, randomized, open-label, parallel controlled trial. A total of 36 participants with T2DM and MASLD (defined by MRI-PDFF ≥10%) will be randomized in a 1:1 ratio to receive either once-daily iGlarLixi or iGlar, both in combination with metformin, for 12 weeks. The primary outcome is the change in liver fat content assessed by magnetic resonance imaging proton density fat fraction (MRI-PDFF) from baseline to week 12. Key secondary outcomes include changes in liver enzymes, liver inflammation, fibrosis indices (assessed by transient elastography and FIB-4 index), body composition (weight, BMI, waist circumference, waist-to-hip ratio, and visceral fat area), glycemic control (HbA1c, fasting and postprandial glucose), insulin function, lipid profiles, and uric acid. Safety assessments will include monitoring of hypoglycemic events, gastrointestinal adverse events, and other adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Type 2 Diabetes Mellitus.
2. Diagnosis of MASLD with liver fat content defined by MRI-PDFF ≥ 10%.
3. HbA1c ≥ 9.0% at screening.
4. Body Mass Index (BMI) between 25.0 and 35.0 kg/m², with stable weight (change < 10% in the past 3 months).
5. Stable antidiabetic regimen for at least 3 months prior to screening.

Exclusion Criteria:

* 1. History of excessive alcohol consumption (≥210 g/week for men, ≥140 g/week for women).

  2. Other known causes of chronic liver disease (e.g., viral hepatitis, autoimmune hepatitis, Wilson's disease, hemochromatosis).

  3. Use of medications known to affect liver fat content (e.g., thiazolidinediones, SGLT2 inhibitors, GLP-1 receptor agonists, systemic corticosteroids) within 3 months prior to screening.

  4. Presence of acute infections or diabetic acute complications (e.g., ketoacidosis, hyperosmolar state) within 2 weeks prior to screening.

  5. History of pancreatitis or elevated amylase/lipase > 3 times the upper limit of normal (ULN).

  6. Significant liver impairment (ALT or AST > 3 × ULN). 7. Moderate to severe renal impairment (eGFR < 60 mL/min/1.73m²). 8. Congestive heart failure (NYHA class III-IV). 9. Personal or family history of medullary thyroid carcinoma (MTC) or Multiple Endocrine Neoplasia syndrome type 2 (MEN-2).

  10. Severe gastrointestinal disease. 11. Contraindications to MRI examination. 12. Pregnancy or lactation. 13. Participation in another investigational drug study within 6 months prior to enrollment.

  14. Known hypersensitivity to the study drugs or their excipients.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-03-29 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes of liver fat content | Baseline, 12 weeks
  The changes of liver fat content were measured by MRI-PDFF

SECONDARY OUTCOMES:
Changes of liver transaminase | Baseline, 12 weeks
  The changes of liver transaminase were measured by ALT, AST, γ-GGT.
Changes of liver inflammation index | Baseline, 12 weeks
  The changes of liver inflammation index were measured by TE.
Changes of liver stiffness measurement | Baseline, 12 weeks
  The changes of liver stiffness measurement were measured by MRE and VCTE.
Changes of FIB-4 index | Baseline, 12 weeks
  The changes of liver fibrosis can be measured by FIB-4 index.
Changes of body weight | Baseline, 12 weeks
  The changes of body weight were measured by InBody-770 equipment.
Changes of body fat | Baseline, 12 weeks
  The changes of body fat were measured by InBody-770 equipment.
Changes of muscle mass | Baseline, 12 weeks
  The changes of muscle mass were measured by InBody-770 equipment.
Changes of HbA1c | Baseline, 12 weeks
  The changes of glucose metabolism indexes were measured by HbA1c.
Changes of plasma glucose | Baseline, 12 weeks
  The changes of glucose metabolism indexes were measured by fasting plasma glucose and 2-h postprandial plasma glucose.
Changes of C-peptide | Baseline, 12 weeks
  The changes of glucose metabolism indexes were measured by fasting C-peptide and 2-h postprandial C-peptide.
Changes of lipid metabolism indexes | Baseline, 12 weeks
  The changes of lipid metabolism indexes were measured by triglyceride, total cholesterol, high-density and low-density lipoprotein-cholesterol.

OTHER OUTCOMES:
Incidence of Hypoglycemic Events | From Baseline to Week 12
  The number and percentage of participants experiencing at least one hypoglycemic event, categorized by severity, will be assessed and compared between treatment groups.
Incidence of other adverse events | From Baseline to Week 12
  All adverse events (AEs) will be recorded and summarized, with particular focus on gastrointestinal adverse events (GIAEs) and other specified events. The following data will be collected: the number and percentage of patients with GIAEs, including the type (nausea, vomiting, diarrhea), grading (per CTCAE v5.0), severity, and relationship to the study drug; the number and percentage of patients with other AEs (including allergic reactions, major adverse cardiovascular events [MACE], and pancreatic events).

CONTACTS AND LOCATIONS:
Overall Officials: Yan Bi, Study Director — Department of Endocrinology, the Affiliated Drum Tower Hospital of Nanjing University Medical School
Locations (1):
- Department of Endocrinology, the Affiliated Drum Tower Hospital of Nanjing University Medical School, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No